CLINICAL TRIAL: NCT00610207
Title: Treatment of Crohn's Fistula Using a Porcine Intestine Submucosa Graft (SurgiSIS AFP)
Brief Title: Treatment of Crohn's Fistula Using a Porcine Intestine Submucosa Graft
Acronym: SurgiSIS AFP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped early due to staffing changes at the site.
Sponsor: Cook Group Incorporated (Industry)
Collaborators: Cook Biotech Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-002
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2012-03

CONDITIONS: Anal Fistula; Crohn's Disease
Keywords: Anal fistula; fistula in ano; anorectal fistula; Crohn's Disease
MeSH Terms: conditions — Rectal Fistula; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AFP (Experimental): Anal fistula plug placement performed during surgical procedure
  Interventions: Device: Surgisis Biodesign Anal Fistula Plug (SurgiSIS AFP)

INTERVENTIONS:
Device: Surgisis Biodesign Anal Fistula Plug (SurgiSIS AFP) — Surgical placement of the Surgisis AFP is performed under general anesthesia
  Other Names: SurgiSIS Biodesign

SUMMARY:
Healing anal fistulas in Crohn's patients with an anal fistula plug.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the Surgisis anal fistula plug is effective in healing anal fistulas in patients diagnosed with Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with Crohn's Disease
* Patient has a chronically draining anal fistula of Crohn's origin
* Patient is 18 years old or older
* Patient has signed an informed consent

Exclusion Criteria:

* Patient is pregnant or lactating
* Patient has peri-anal drainage with originates from outside the anorectal tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Moore, MD, Principal Investigator — Colon & Rectal Surgeons of Southern California, Mt. Sinai
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mount Sinai Medical Center, New York, New York
  - Univeristy Hospitals Medical Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Biodesign® Anal Fistula Plug: Biodesign is a bioprosthetic material derived from porcine small intestinal submucosa (SIS) that provides mechanical integrity while acting as a scaffold to guide tissue incorporation.
  Three single tract fistula patients were lost to follow-up and were excluded from the analysis.
Period: Overall Study
Arm/Group | Biodesign® Anal Fistula Plug
Started | 21
Completed | 18
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Biodesign® Anal Fistula Plug
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] — Three single-tract fistula patients were lost to follow-up and were excluded from the analysis on age.
  years | 40.2 [22 to 69]
Sex: Female, Male [Count of Participants; unit: Participants] — Three single-tract fistula patients were lost to follow-up and were excluded from the analysis on gender.
  Participants
    Female | 9
    Male | 9
Height [Mean (Full Range); unit: inches] — Three single-tract fistula patients were lost to follow-up and were excluded from the analysis on height.
  inches | 66 [59 to 72]
Weight [Mean (Full Range); unit: pounds] — Three single-tract fistula patients were lost to follow-up and were excluded from the analysis on weight.
  pounds | 148 [85 to 208]
Body Mass Index [Mean (Full Range); unit: kg/m^2] — Three single-tract fistula patients were lost to follow-up and were excluded from the analysis on body mass index.
  kg/m^2 | 24 [14 to 37]

OUTCOME MEASURES:

1. Primary Outcome: Fistula Closure (Patient Based)
Description: Fistula closure is defined as absence of drainage at the external fistula opening.
Time Frame: 12 months
Population: Three single tract fistula patients were lost to follow-up and were excluded from the analysis.
Measure: Number; unit: participants
Arm/Group | Biodesign® Anal Fistula Plug
Number analyzed (Participants) | 18
participants | 10

2. Primary Outcome: Fistula Closure (Tract Based)
Description: Fistula closure is defined as absence of drainage at the external fistula opening.
  An anorectal fistula is an inflammatory tract or connection between the epithelialized surface of the anal canal and most frequently, the perianal skin or perineum. It is possible to have multiple fistula tracts present on a patient.
Time Frame: 12 months
Population: Three single tract fistula patients were lost to follow-up and were excluded from the analysis.
Measure: Number; unit: tracts
Units Other Than Participants: tracts
Arm/Group | Biodesign® Anal Fistula Plug
Number analyzed (Participants) | 18
Number analyzed (tracts) | 25
tracts | 17

ADVERSE EVENTS:
Time Frame: 12 months
Description: Three single-tract fistula patients were lost to follow-up and were excluded from the analysis.
Arm/Group | Biodesign® Anal Fistula Plug
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
Early termination did lead to small patient numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less